CLINICAL TRIAL: NCT07079371
Title: Assessment of the Effect of Micellar Solution on Measures of Skin Barrier Function
Brief Title: Micellar Water and the Skin Barrier: Comparing Rinsing vs. Non-Rinsing Application
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2181-198-03-04-25-0065
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Effects of Micellar Water Application on Skin Barrier Integrity, Hydration, and Erythema in Healthy Skin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micellar Water Application Without Rinsing (Experimental): Participants apply micellar water to the forehead once daily and leave it on the skin without rinsing. Skin barrier function is assessed before and after 21 days of application.
  Interventions: Procedure: Micellar Water Application (No Rinse)
- Micellar Water Application With Rinsing (Experimental): Participants apply micellar water to the forehead once daily and rinse it off after application. Skin barrier function is assessed before and after 21 days of application.
  Interventions: Procedure: Micellar Water Application (With Rinse)

INTERVENTIONS:
Procedure: Micellar Water Application (No Rinse) — Participants apply micellar water to the forehead once daily and leave it on the skin without rinsing for 21 days.
  Arms: Micellar Water Application Without Rinsing
Procedure: Micellar Water Application (With Rinse) — Participants apply micellar water to the forehead once daily and rinse it off after application for 21 days.
  Arms: Micellar Water Application With Rinsing

SUMMARY:
The goal of this clinical trial is to assess how micellar water affects the skin barrier in healthy adult volunteers. The main questions it aims to answer are:

* Does leaving micellar water on the skin affect skin barrier function differently than rinsing it off?
* Are there measurable differences in transepidermal water loss (TEWL), skin hydration, and erythema between the two application methods?

Researchers will compare the effects of micellar water left on the skin versus rinsed off after application.

Participants will:

* Be randomly assigned to one of two groups
* Apply micellar water to their forehead once daily for 21 days
* Either leave the micellar water on or rinse it off, depending on their group
* Undergo non-invasive measurements of TEWL, skin hydration, and erythema before and after the intervention

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 18 years and older. Willingness and ability to comply with study procedures. Signed informed consent indicating understanding of study participation, rights, and potential risks and benefits. No current skin diseases or conditions at the test site. Ability to attend all study visits and follow instructions

Exclusion Criteria:

* Participants with skin diseases, skin cancers, or sun damage at the test site will be excluded. Use of immunomodulators, corticosteroids, or antihistamines within 30 days prior to the study start is exclusionary. Application of emollient creams within 3 days before the trial is not permitted. Other exclusion criteria include protocol non-compliance, excessive exposure to natural or artificial ultraviolet radiation, pregnancy or lactation, history of vitiligo, melasma, or other hyperpigmentation or photosensitive disorders, immunosuppression, and allergy to any ingredient of the micellar solution used in the intervention. Before starting the study, participants will be asked if they have ever experienced adverse reactions to any components of the micellar solution.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in TransEpidermal Water Loss (TEWL) | Four measurements total: one at baseline (before application), and one at the start of each week during the 3-week intervention (Days 0, 7, 14, and 21).
  Measurement of transepidermal water loss on the forehead to assess skin barrier function.
Change in Skin Hydration | Four measurements total: one at baseline (before application), and one at the start of each week during the 3-week intervention (Days 0, 7, 14, and 21).
  Measurement of skin hydration levels on the forehead before and after micellar water application.
Change in Erythema | Four measurements total: one at baseline (before application), and one at the start of each week during the 3-week intervention (Days 0, 7, 14, and 21).
  Assessment of skin redness (erythema) on the forehead before and after of micellar water application.

CONTACTS AND LOCATIONS:
Locations (1):
- Univerity of Split School of Medicine, Split, Croatia